CLINICAL TRIAL: NCT06887179
Title: The Role of Point-of-Care Ultrasound in the Management of Chronic Heart Failure
Brief Title: Point-of-Care Ultrasound in Chronic Heart Failure
Acronym: POCUS-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: University Hospital Brno (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POCUS-HF-FNBrno
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
Keywords: Heart failure; Diuretic therapy; Congestion; Point-of-Care Ultrasound
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study is a randomized, open-label, intention-to-treat, prospective clinical trial.
  It compares ambulatory patients following hospitalization for heart failure in the standard care treatment arm with the intervention arm treated according to the HF-focused POCUS results done by the treating physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): * Echocardiography in index hospitalization (left ventricle ejection fraction, E/e' ratio, LAVi, TAPSE, peak systolic tricuspid annular velocity, peak tricuspid regurgitation velocity, estimated pulmonary artery systolic pressure)
  * Mini-Mental State Examination in index hospitalization in 65 years and older
  * Clinical examination, blood pressure, heart rate, oxygen saturation, ECG, height, weight, BMI, NYHA on every visit
  * KCCQ in first week visit and 12 months visit
  * Blood tests:
    * NT-proBNP in index hospitalization and 12 months visit
    * blood count, urea, creatinine, glycaemia and electrolytes on every visit
  * HF focused POCUS on every visit
  Interventions: Procedure: HF focused POCUS
- Standard care arm (Active Comparator): * Echocardiography in index hospitalization (left ventricle ejection fraction, E/e' ratio, LAVi, TAPSE, peak systolic tricuspid annular velocity, peak tricuspid regurgitation velocity, estimated pulmonary artery systolic pressure)
  * Mini-Mental State Examination in index hospitalization in 65 years and older
  * Clinical examination, blood pressure, heart rate, oxygen saturation, ECG, height, weight, BMI, NYHA on every visit
  * KCCQ in first-week visit and 12 months visit
  * Blood tests:
    * NT-proBNP in index hospitalization and on every scheduled visit
    * blood count, urea, creatinine, glycaemia and electrolytes on every visit
  Interventions: Procedure: Standard Care (in control arm)

INTERVENTIONS:
Procedure: HF focused POCUS — * POCUS findings guide diuretic therapy adjustments by treating physicians
  * POCUS is performed with handheld device Vscan air SL® or Vscan extend®, GE Healthcare.
  * Sector probe and abdominal preset are used. Only B-mode is used.
  * The image depth is 15 cm or more to evaluate the structures sufficiently.
  * Patient position is supine or semirecumbent. For the pleural effusion exam, the preferred position is sitting.
    1. Lungs: Assessment of B-lines in midclavicular and midaxillary zones.
    2. Pleural Effusion
    3. Inferior Vena Cava
    4. Ascites
  Arms: Intervention Arm
Procedure: Standard Care (in control arm) — Standard care assessment with NT-proBNP on every scheduled visit.
  Arms: Standard care arm

SUMMARY:
This study aims to determine whether Point-of-Care Ultrasound (POCUS)-guided treatment is non-inferior to standard NT-proBNP-based care in ambulatory patients following hospitalization for heart failure (HF) over a 12-month follow-up period.

DETAILED DESCRIPTION:
Although ultrasound machines are routinely available in ambulatory settings these days, assessing congestion with POCUS during regular visits is not yet established as a standard of care for HF patients. Accurate assessment of congestion is a cornerstone in managing HF since congestion is a major driver of symptoms, hospitalizations, and adverse outcomes. Current standard methods for congestion assessment include clinical examination, laboratory markers such as NT-proBNP, chest X-ray, and sometimes invasive hemodynamic monitoring. However, these approaches have limitations: clinical signs can be subjective, NT-proBNP levels may be influenced by non-cardiac factors, and invasive monitoring is not feasible for routine outpatient use. Chest X-ray bears the risk of irradiation and is more time and money-consuming than bedside tools.

POCUS has emerged as a promising tool for real-time congestion assessment. It allows for direct visualization of pulmonary and systemic congestion, providing rapid bedside insights into the patient's volume status (9). Despite its advantages, POCUS is not yet widely implemented in routine HF ambulatory management, primarily due to the lack of standardized protocols with sufficient evidence.

This study evaluates whether an HF-focused POCUS protocol can enhance congestion assessment in ambulatory HF patients following hospitalization. During a follow-up period of 12 months, they will be regularly examined clinically and with standard laboratory tests. HF-focused POCUS will be performed in the interventional arm instead of standard NT-proBNP testing. For the sake of simplicity and practicality of the examination, a handheld ultrasound device (GE Healthcare Vscan Air SL® or Vscan Extend®) with only a sector probe in B-mode will be employed.

The HF-focused POCUS examination includes several predefined components. Lung assessment to detect pulmonary congestion. Pleural assessment to detect congestion with effusion. The inferior vena cava assessment is used to estimate central venous pressure. The presence of ascites is evaluated by scanning the hepatorenal space and right paracolic gutter for signs of fluid accumulation.

The HF-focused POCUS is performed by treating physicians, allowing immediate diuretic therapy adjustments based on the results. The hypothesis is that HF-focused POCUS can enable more precise diuretic titration, potentially reducing adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients after hospitalization for acute heart failure (AHF)
* Symptoms (shortness of breath, oedema, decreased exercise tolerance, increase in abdominal circumference)
* Clinical signs (jugular vein distention, hepatojugular reflux, third heart sound, wet lung crackles, pitting oedema) or signs of congestion on CT, X-ray or ultrasound
* NT-proBNP >450 pg/mL <55 years old, >900 pg/mL 55-75 years old, >1800 pg/mL >75 years old
* Increase in oral diuretic therapy or need for IV diuretics

Exclusion Criteria:

* pregnancy or lactation
* under 18 years of age,
* current AHF due to a transient cause (Takotsubo syndrome, neurogenic myocardial stunning, septic cardiomyopathy, cardiac tamponade, pulmonary embolism with acute cor pulmonale, thyrotoxicosis, bradycardia <40/min)
* planned surgical treatment of the HF cause, CRT implantation or valvular repair ≤ 30 days ago, STEMI or coronary angiography with PCI or CABG ≤ 30 days ago, untreated AV block III. and II. degree type 2, planned or previous heart transplantation, myocarditis ≤ 6 months ago, complex congenital heart disease, cardiac amyloidosis, hypertrophic and restrictive cardiomyopathy, constrictive pericarditis
* BMI over 40 kg/m2, cognitive deficit with MMSE <18 points, life expectancy < 12 months, progressive oncological disease, chronic liver failure Child-Pugh C, chronic kidney disease with eGFR <0.25 ml/s
* current participation in another study or relative of investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome | 12 months
  The primary outcome is a composite of urgent visits, hospitalization for worsening HF and death from any cause. We defined an urgent visit for worsening HF as an unscheduled visit because of signs and/or symptoms of worsening HF that require IV diuretic treatment or a diuretic increase with a hospital stay of less than 24 hours. Hospitalization for worsening HF is defined as a stay in hospital for more than 24 hours because of signs and/or symptoms of worsening HF.

SECONDARY OUTCOMES:
The number of all AHF hospitalizations | 12 months
  The total number of all AHF hospitalizations
The number of other unplanned hospitalizations | 12 months
  The total number of other unplanned hospitalizations
The number of all unscheduled visits for any cause | 12 months
  The total number of all unscheduled visits for any cause
The number of extra visits beyond the protocol schedule for HF treatment | 12 months
  The total number of extra visits beyond the protocol schedule for HF treatment
The change in NT-proBNP | 12 months
  The change in NT-proBNP (ng/l)
The change in eGFR | 12 months
  The change in eGFR (ml/s/1,73m2)
The change in Kansas City Cardiomyopathy Questionnaire | 12 months
  The change in KCCQ (points). It is scored from 0 to 100 with higher scores indicating better health status.
The number of performed chest X-rays | 12 months
  The total number of performed chest X-rays
The number of drainage procedures for fluidothorax or ascites. | 12 months
  The total number of drainage procedures for fluidothorax or ascites.
Safety outcome | 12 months
  Diuretics-related decrease in eGFR >50% (with signs of hypovolemia) compared to the 1st-week visit value; the level of hypokalemia <3.5 mmol/L (the number of patients having hypokalemia <3.5 mmol/L).
The level of hypokalemia <3.5 mmol/L | 12 months
  The number of patients having hypokalemia <3.5 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Ludka, Prof., Study Chair — University Hospital Brno; Ondrej Ludka, Prof., Study Director — University Hospital Brno; Adam Koudelka, MD, Principal Investigator — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No